CLINICAL TRIAL: NCT00135746
Title: Effects of Transdermal Nicotine on Tobacco Withdrawal and the Effects of Smoking in Men and Women
Brief Title: Examining the Effectiveness of the Nicotine Patch in Male and Female Smokers - 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Thomas Eissenberg, Virginia Commonwealth University
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-11082-2; R01-11082-2; DPMC
Record Dates: First submitted 2005-08-23; First posted 2005-08-26 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2015-10

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Drug: nicotine transdermal system

SUMMARY:
Treatment studies have demonstrated that current smoking cessation techniques are less effective for women. The purpose of this study is to determine the role that gender plays on the effectiveness of nicotine replacement therapy. This may lead to improved cessation interventions for all smokers, particularly women.

DETAILED DESCRIPTION:
Currently, about 70 percent of smokers who try to quit by using smoking cessation treatments are unsuccessful. Treatment studies have demonstrated that current smoking cessation techniques are less effective for women. There is no clear explanation for this difference, but it may involve a differential response to nicotine replacement treatments (NRTs) and/or smoking-related stimuli. For women, NRT may be less effective at suppressing withdrawal or blunting the effects of smoking during a quit attempt. Women may also be more sensitive to smoking-related stimuli, such as the taste, sight, and smell of smoke. Tailoring treatment to the separate needs of subgroups, such as men and women, may produce better outcomes. The purpose of this study is to assess the influence of gender on the effectiveness of transdermal nicotine treatment in a group of male and female smokers.

Participants in this double-blind, dose-comparison study will complete separate sessions in a random order.

Each session will last approximately 6.5 hours and will correspond to a specific transdermal patch dose (0, 7, 14, or 21 mg). Objectively verified cigarette abstinence will be required before each session. Sessions will occur at least 48 hours apart to avoid carryover. Cognitive, behavioral, subjective, and physiological measures will occur during study visits. Specifically, the NRT dose response to tobacco suppression and cigarette blunting effects will be compared in women and men.

ELIGIBILITY:
Inclusion Criteria:

* Daily cigarette use of 15 or more cigarettes for at least 2 years
* Screening CO level of or greater than 15 ppm
* Normal or corrected-to-normal vision
* Willing to abstain from tobacco products for 8 or more hours prior to testing

Exclusion Criteria:

* History of chronic health problems or psychiatric conditions
* History of cardiovascular disease, low or high blood pressure, seizures, head injuries requiring hospital care, peptic ulcer, or diabetes
* Pregnancy (tested by urinalysis)
* Scores greater than 17 on the Beck Depression Inventory
* Lack of a high school degree or GED

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2004-05; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Subjective effects
Cognitive performance
Physiologic measures
Smoking Behavior
Plasma Nicotine

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eissenberg, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Behavioral Pharmacolgy Research Laboratory, Richmond, Virginia, United States